CLINICAL TRIAL: NCT06753136
Title: Treatment of Visceral Localizations With Electrochemotherapy in Patients With Primary Visceral Tumors and/or Secondary Visceral Localizations, of Any Histotype: Monocenter, Single Arm, Clinical Investigation
Brief Title: Electrochemotherapy (ECT) in Patients With Primary Visceral Tumors and/or Secondary Visceral Localizations, of Any Histotype
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: IGEA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-VL-01-2024-ECT
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Primary Visceral Tumors of Any Histotype; Visceral Lesions; Liver Cancer; Liver Metastasis Colon Cancer; Melanoma; Primary Pancreatic Tumor; Retroperitoneal Sarcoma; Abdominal and/or Peritoneal Localizations; Merkel Cell Carcinoma; Squamous Cell Carcinoma; Secondary Visceral Localizations of Any Histotype; Non-melanoma Skin Cancer
Keywords: electrochemotherapy; visceral lesions; Laparoscopic procedure; Laparotomic procedure; Percutaneous procedure; bleomycin; medical device
MeSH Terms: conditions — Liver Neoplasms; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Squamous Cell | interventions — Administration, Cutaneous; Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- electrochemotherapy (Experimental): Patients who meet the inclusion criteria will undergo percutaneous, laparoscopic or laparotomy lesion electrochemotherapy within 30 days from the time of obtaining informed consent for study participation (T0), during pre-surgery visit.The ECT will be performed in accordance with the Standard Operating Procedures (SOPs).During the first month after treatment, the patient's response will be assessed every 2 weeks, and thereafter, once a month for a total of 12 months.
  Interventions: Device: percutaneous, laparoscopic or laparotomy lesion electrochemotherapy

INTERVENTIONS:
Device: percutaneous, laparoscopic or laparotomy lesion electrochemotherapy — All patients will receive Bleomycin intravenously with a dosage of 15.000 IU/m2. After a drug distribution time of 8 minutes, the lesions will be electroporated using the Cliniporator (IGEA S.P.A., Carpi, Italy), applying special handpieces depending on the route used: laparoscopic electrode, flexible and expandable for the laparoscopic procedure, linear or hexagonal electrode for laparotomy surgical access, variable geometry electrode for percutaneous access. The ECT procedure must be completed within 40 minutes.

SUMMARY:
This is an monocenter, single arm, clinical investigation that evaluate the impact of the method on the objective response rate (ORR) of visceral lesions undergoing electrochemotherapy. Electrochemotherapy is a well-defined method for the treatment of cutaneous and subcutaneous metastases of different tumor histotypes.

Although still limited, the various experiences in the treatment of visceral localizations, particularly in liver metastases from colorectal cancer are promising and show that electrochemotherapy is a safe treatment, even in the case of lesions near large vessels or nerves. The investigators therefore propose a clinical investigation with a Medical Device according to EU Regulation 745/2017, using electrochemotherapy (Cliniporator) with bleomycin for the treatment of visceral, primary or secondary, unresectable localizations, with percutaneous or intraoperative technique (laparoscopic or laparotomy), as needed.

DETAILED DESCRIPTION:
This is a single-center clinical investigation with the enrollment of at least 24 patients with visceral, primary or secondary localizations, of any histotype, with particular reference to liver cancer, liver metastases from colorectal cancer and melanoma, primary pancreatic tumors, retroperitoneal sarcomas, abdominal and/or peritoneal localizations from melanoma and non-melanoma skin cancer (Merkel cell carcinoma, Squamous cell ca).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female ≥ 18 years
* Ability to understand the proposed treatment and express an informed acceptance by signing the informed consent
* Diagnosis of primary and/or secondary visceral localizations of any histotype
* Patients who are not eligible for standard curative procedures

Exclusion Criteria:

* Absolute contraindications to invasive procedures
* Concomitant presence of brain, lung, bone metastases
* Uncorrectable coagulation changes
* Bleomycin allergy
* Absolute contraindications to taking Bleomycin
* Poor respiratory function or pulmonary fibrosis
* Acute lung infections
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary objective and endpoint | through study completion, an average of 5 year
  Evaluate the impact of the method on the objective response rate (ORR) of visceral lesions undergoing electrochemotherapy. ORR is defined as the proportion of patients, out of the total enrolled subjects, who achieved a complete response (CR) or partial response (PR) response, based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Determination of radiological response will be based on the assessment reported by the investigator. Radiological responses will be assessed every 8 weeks starting with cycle 1 day 1 of treatment until disease progression, withdrawal of consent, or death for any reason, whichever occurs first.

SECONDARY OUTCOMES:
Secondary objective and endpoints | through study completion, an average of 5 year
  Evaluate the conversion rate of "unresectable disease" to "resectable disease" after ECT treatment. The conversion from "unresectable disease" to "resectable disease" is defined by the number of patients, declared inoperable with the intent of surgical radicality due to the extent of the disease and/or the involvement of non-removable structures and who become operable for surgery with the intent of radical excision following response after an electrochemotherapy treatment.
Secondary objective and endpoints | through study completion, an average of 5 year
  Assess progression-free time (PFS). Progression-free survival (PFS) is defined as the time from study enrollment to the first documentation of objective disease progression or death due to any cause, whichever occurs first. Documentation of disease progression is defined according to RECIST v1.1 criteria, based on investigator assessment. PFS will be censored at the time of the last tumor evaluation documenting the absence of progression for patients who are alive and progression-free at the time of analysis. Live patients who have no tumor assessments after baseline will have time to the censored event on the date of study enrollment.
Secondary objective and endpoints | through study completion, an average of 5 year
  Assess overall survival (OS). Overall survival (OS) is defined as the time (quantified in months) from enrollment in the study to the date of the subject's death from any cause. For subjects living at the end of the study, the last follow-up date will be considered.
Secondary objective and endpoints | through study completion, an average of 5 year
  Evaluate the toxicity of electrochemotherapy treatment (ECT). Overall toxicity rate is defined as the proportion of patients, among those who received at least one dose of treatment, who experienced grade 3-4 adverse events, according to NCI CTCAE v5.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided